CLINICAL TRIAL: NCT02784015
Title: Response-based Treatment for Children With Unresectable Localized Soft Tissue Sarcomas
Brief Title: Response Based Treatment for Children With Unresectable Localized Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-07-115
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Unresectable Localized Soft Tissue Sarcoma
MeSH Terms: interventions — Cisplatin; Etoposide; Doxorubicin; Cyclophosphamide; Ifosfamide; Carboplatin; Radiotherapy; Thiotepa; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Unresectable localized soft tissue sarcoma (Experimental): 1. Six cycles of chemotherapy with cisplatin, etoposide, doxorubicin, cyclophosphamide (CEDC) and ifosfamide, carboplatin, etoposide (ICE) regimen.
  2. Surgery, if possible
  3. Concurrent chemoradiotherapy according to the treatment response (necrosis rate, tumor volume reduction, and residual FDG uptake in PET scan)
  4. Tandem high dose chemotherapy (HDCT) and autologous stem cell transplantation, if there are still residual tumors after 9 cycle of chemotherapy, surgery, and radiotherapy.
     * 1st HDCT: carboplatin, thiotepa, etoposide
     * 2nd HDCT: cyclophosphamide, melphalan
  Interventions: Drug: Cisplatin; Drug: Etoposide; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Ifosfamide; Drug: Carboplatin; Radiation: Radiotherapy; Drug: Thiotepa; Drug: Melphalan

INTERVENTIONS:
Drug: Cisplatin
Drug: Etoposide
Drug: Doxorubicin
Drug: Cyclophosphamide
Drug: Ifosfamide
Drug: Carboplatin
Radiation: Radiotherapy
Drug: Thiotepa
Drug: Melphalan

SUMMARY:
To evaluate the treatment outcome of unresectable soft tissue sarcoma using response based treatment

DETAILED DESCRIPTION:
Response after initial chemotherapy is one of the important prognostic factor in many cancers. In this study, treatment will be tailored according to the treatment responses which are assessed by tumor volume reduction, necrosis rate or residual fludeoxyglucose (FDG) uptake in positron emission tomography (PET) scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable localized high grade soft tissue sarcoma

Exclusion Criteria:

* Patients with organ dysfunction (ejection fraction, liver function test, creatinine > CTCAE grade 2)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Rate of event free survival | Up to 3 years

SECONDARY OUTCOMES:
Rate of adverse events | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea